CLINICAL TRIAL: NCT04792177
Title: SHER 2: Internet-delivered Emotion Regulation Skills Training for Sexual Health: a Randomized Controlled Trial
Brief Title: Internet-based Emotion Regulation Intervention for Sexual Health
Acronym: SHER2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luxembourg (Other)
Collaborators: Luxembourg National Research Fund (FNR) (Unknown); Linkoeping University (Other Government); University of Lausanne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHER 20-029
Record Dates: First submitted 2021-01-29; First posted 2021-03-10 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Sexual Dysfunction; Sexual Dysfunctions, Psychological
Keywords: internet intervention; emotion regulation; sexual health
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups for the duration of the study. 50% of participants will be assigned to the intervention group while the other 50% will be assign to a waitlist control condition. The waitlist group will have access to the intervention after 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Emotion regulation skills training group
  Interventions: Behavioral: Emotion regulation skills training
- waitlist control group (No Intervention): The control group will not receive any intervention during the trial but will be offered the same treatment at the end of the six-months follow-up assessment.

INTERVENTIONS:
Behavioral: Emotion regulation skills training — The intervention will involve an online emotion-regulation skills training for individuals with sexual problems. It will last for 8 weeks, encompassing psycho-educational and emotion-regulation skills components. Every week participants will gain access to a different intervention module of the training, containing videos, presentation slides, written support material and a recommendation of activities to be completed until the following week of training. Participants are expected to dedicate 30 minutes to one hour per week to complete each module.
  Arms: Intervention group

SUMMARY:
Introduction: Emotion regulation difficulties have been associated with mental disorders and sexual dysfunctions. Traditional face-to-face transdiagnostic emotion regulation interventions have shown positive results for emotional and personality disorders. Only recently have the effects of these interventions on sexual health started to be investigated. Internet-delivered psychological interventions have several advantages over face-to-face interventions, such as cost-effectiveness, accessibility and suitability for people who experience shame because of their stigmatized problematic behaviors and those who avoid seeking help. The aims of the SHER 2 study are: a) determine the efficacy of an Internet-based emotion regulation intervention for sexual health and sexual satisfaction, and; b) explore the effects of the intervention on (1) emotion regulation skills; (2) mental health; (3) sexual self-perception.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years of age,
* fluent in Brazilian Portuguese,
* self-reported sexual problems, assessed in men by a score of < 21 on the International Index Erectile Function (IIEF) and in women by a score of < 26 on the Female Sexual Function Index (FSFI),
* in a stable relationship for at least the preceding 3 months.

Exclusion Criteria:

* medical conditions that can interfere with the outcomes of the intervention, e.g., diabetes, cancer, cardiovascular problems,
* ongoing psychotherapy.
* no sexual activity in the previous 4 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Female Sexual Function Index (FSFI) at 6 months | baseline, 2 months after baseline (end of intervention), 8 months after baseline (follow-up)
  this is a 19-item questionnaire for the assessment of sexual functioning in women in domains of sexual functioning (e.g., sexual arousal, orgasm, satisfaction, pain). Answers are provided using a 5-point Likert scale.
Change in International Index of Erectile Function (IIEF)at 6 months | baseline, 2 months after baseline (end of intervention), 8 months after baseline (follow-up)
  The IIEF is 15-item, self-administered questionnaire for assessing sexual functioning in men. Answers are given on a 6-point Likert scale. The IIEF encompasses five different domains of sexual functioning: erectile function, orgasm function, sexual desire, intercourse satisfaction and overall satisfaction.
Change in Sexual Quotient (QS) at 6 months | baseline, 2 months after baseline (end of intervention), 8 months after baseline (follow-up)
  The QS is a brief and comprehensive tool composed of 10-questions, which are answered on a scale from 0 (never) to 5 (always). It addresses general sexual function, and stages of the sexual response cycle (desire, arousal, orgasm) and sexual satisfaction.

SECONDARY OUTCOMES:
Sexual Modes Questionnaire (SMQ) - Automatic Thoughts subscale | baseline, 2 months after baseline (end of intervention), 8 months after baseline (follow-up)
  This self-report scale consists of 30 items in the male version, and 33 items in the female version. Respondents are asked to rate the frequency (from 1 [never] to 5 [always]) with which they have experienced specific automatic thoughts during sexual activity.
Sexual Self-Schema Scale (SSSS). | baseline, 2 months after baseline (end of intervention), 8 months after baseline (follow-up)
  consists of 30 items assessing respondents' perception of themselves as a sexual person compared to others of the same gender and age. Answers are provided using a 5- point Likert scale ranging from 1 (not at all descriptive of me) to 5 (very much descriptive of me).
Patient Health Questionnaire-9 (PHQ-9) | baseline, 2 months after baseline (end of intervention), 8 months after baseline (follow-up)
  A 9-item self-report measure used to assess symptoms of depression.
General Anxiety Disorder - 7 (GAD-7) | baseline, 2 months after baseline (end of intervention), 8 months after baseline (follow-up)
  A 7-item self-report measure used to assess symptoms of anxiety.
the Difficulties in Emotion Regulation Scale (DERS) | baseline, 2 months after baseline (end of intervention), 8 months after baseline (follow-up)
  The DERS assesses several facets of emotion regulation, including difficulties relevant to an individual's (a) acceptance of emotional responses, (b) ability to engage in goal-directed behaviour under distress, (c) ability to control impulsive behaviours when distressed, (d) access to emotion regulation strategies, and (e) emotional clarity. Participants rate their degree of agreement with each statement on a scale from 1 (almost never; 0 to 10 percent) to 5 (almost always; 91 to 100 percent).

CONTACTS AND LOCATIONS:
Overall Officials: Claus Vögele, Prof. Dr, Principal Investigator — Head of Department Department of Behavioural and Cognitive Sciences
Locations (1):
- University of Luxembourg, Esch-sur-Alzette, Luxembourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jobim Fischer V, Rossato Holz M, Billieux J, Andersson G, Vogele C. Web-Based Emotion Regulation Training for Sexual Health: Randomized Controlled Trial. JMIR Form Res. 2024 Apr 3;8:e50850. doi: 10.2196/50850. PMID 38568720
- See also: Related Info — http://treps.iterapi.se